CLINICAL TRIAL: NCT06284668
Title: Esketamine vs Remimazolam for Postoperative Sleep Disturbance and Anxiety in Patients Undergoing Oocyte Retrieval
Brief Title: Esketamine vs Remimazolam for Postoperative Sleep Disturbance and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang027
Record Dates: First submitted 2024-02-01; First posted 2024-02-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disturbance
Keywords: Esketamine; Remimazolam; oocyte retrieval
MeSH Terms: conditions — Parasomnias | interventions — Saline Solution; Esketamine; remimazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group of patients undergoing oocyte retrieval with normal saline (Placebo Comparator): Patients undergoing oocyte retrieval were given 5ml 0.9% saline before anesthesia and surgery
  Interventions: Drug: normal Saline
- Group of patients undergoing oocyte retrieval with esketamine (Active Comparator): Patients undergoing oocyte retrieval were given esketamine 0.2mg/kg before anesthesia and surgery
  Interventions: Drug: Esketamine
- Group of patients undergoing oocyte retrieval with remimazolam (Active Comparator): Patients undergoing oocyte retrieval were given remimazolam 0.2mg/kg before anesthesia and surgery
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: normal Saline — Patients undergoing oocyte retrieval were given 5ml 0.9% saline before anesthesia and surgery
  Other Names: Group of patients undergoing oocyte retrieval with normal saline
  Arms: Placebo Group of patients undergoing oocyte retrieval with normal saline
Drug: Esketamine — Patients undergoing oocyte retrieval were given esketamine 0.2mg/kg before anesthesia and surgery
  Other Names: Group of patients undergoing oocyte retrieval with esketamine
  Arms: Group of patients undergoing oocyte retrieval with esketamine
Drug: Remimazolam — Patients undergoing oocyte retrieval were given remimazolam 0.2mg/kg before anesthesia and surgery
  Other Names: Group of patients undergoing oocyte retrieval with remimazolam
  Arms: Group of patients undergoing oocyte retrieval with remimazolam

SUMMARY:
To explore and compare the effects of esketamine and remimazolam on postoperative sleep disturbance in patients undergoing oocyte retrieval

DETAILED DESCRIPTION:
Postoperative sleep disturbance (PSD) occur in the form of sleep deprivation, circadian rhythm disturbance, and structural abnormalities, and have a high incidence in patients undergoing surgery. Postoperative sleep disorders can lead to postoperative delirium and cognitive dysfunction, aggravate postoperative acute pain, and delay postoperative recovery.

Benzodiazepines have a certain sedative hypnotic anti-anxiety effect, and remimazolam as a new benzodiazepine, its sedative hypnotic anti-anxiety effect is worthy of further exploration. Esketamine is an N-methyl-D-aspartate(NMDA) receptor antagonist with analgesic and sedative effects, and is widely used in clinical treatment of refractory depression. For patients undergoing surgery, in addition to sedation and analgesia, whether the intraoperative use of esketamine has positive effects on postoperative sleep disturbance is worth exploring.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years old;
2. American society of Aneshesiologists（ASA）physical status classification system is grade I-III;
3. Elective surgery is proposed
4. BMI of 19-30 kg/m2;
5. Patients who agreed to enroll in this study voluntarily

Exclusion Criteria:

1. Those who are known to be allergic to the drug ingredients in this study and their allergic constitution;
2. Allergic history of general anesthesia drugs, opioid drugs, non-steroidal drugs;
3. History of neurological diseases; History of chronic pain; Drug and alcohol addiction; A long history of opioid use; Opiates were given 48 hours before surgery
4. Coronary heart disease, bronchial asthma, severe hypertension, severe blood system dysfunction, liver and kidney function, electrolyte abnormalities;
5. Respiratory insufficiency, respiratory failure;
6. BMI<18 kg/m2 or BMI>30kg/m2;
7. Poor compliance, unable to complete the experiment according to the study plan; Participants who have participated in clinical trials of other drugs within the last 4 weeks;
8. Preoperative Pittsburgh Sleep Quality Index (PSQI) higher than 7
9. Any circumstances deemed unsuitable for inclusion by the researcher for any reason.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative sleep disturbance on the first night after surgery | the first night after surgery
  Patients completed the sleep quality scale(AIS, Athens Insomnia Scale) on the first day after surgery.The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire after the first postoperative night to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.

SECONDARY OUTCOMES:
The incidence of sleep disturbance one day before surgery | one day before surgery
  Patients completed the sleep quality scales(AIS, Athens Insomnia Scale) on the day before surgery.The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia. We asked the patients to fill out this questionnaire on the day before surgery to evaluate patients' preoperative sleep quality. We recorded AIS scores as statistical indicators.
The incidence of postoperative sleep disturbance on the second and third postoperative nights | the second and third nights after surgery
  Patients completed the sleep quality scale(AIS, Athens Insomnia Scale) on the second and third day after surgery.The AIS has a total of 8 items,with scores ranging from 0 to 24 points, and a total score of 6 points or higher indicates a diagnosis of insomnia.We asked the patients to fill out this questionnaire after the second and third postoperative nights to evaluate the changes in sleep quality. We recorded AIS scores as statistical indicators.
Postoperative anxiety | 1 day before surgery ,1 and 2 days after surgery
  Patients completed the anxiety rating scales(HADS-A,Hospital Anxiety and Depression Scale-Anxiety subscale)on the day before surgery.HADS-A consists of 7 items,each question in the questionnaire was scored on a scale of 0-3, and a total score of 8 points or higher is diagnosed as anxiety.And we asked the patients to fill out this questionnaire on the 1 and 2 days after surgery again to evaluate the changes in anxiety. We recorded HADS-A scores as statistical indicators.
Postoperative depression | 1 day before surgery ,1 and 2 days after surgery
  Patients completed the depression rating scales(HADS-D,Hospital Anxiety and Depression Scale-Depression subscale)on the day before surgery.HADS-D consists of 7 items,each question in the questionnaire was scored on a scale of 0-3, and a total score of 8 points or higher is diagnosed as depression.And we asked the patients to fill out this questionnaire on the 1 and 2 days after surgery again to evaluate the changes in depression. We recorded HADS-D scores as statistical indicators.
Pain Score (NRS) | 1 and 2 days after surgery
  The pain score at rest or after movement was evaluated by pain 11-point numerical rating scale (NRS): 0 = no pain, 10 = greatest imaginable pain.
Mean intraoperative blood pressure | Intraoperative
  The mean intraoperative blood pressure was recorded
Oxygen saturation | Intraoperative
  The mean intraoperative oxygen saturation was recorded
Somatokinetic reaction | Intraoperative
  The number of intraoperative body movements was recorded
Operation time | Intraoperative
  The duration of the patient's operation was recorded(up to 24 h)
Duration of anesthesia | Intraoperative
  The patient's duration of anesthesia was recorded(up to 24 h)
Time to walking down | Within1 hour after surgery
  Record the time from waking up to walking down(up to 24 h)
Adverse event | Within 3 days after surgery
  All kinds of adverse events(PONV、hypotension、hypertension,etc) occurred in patients were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, Study Director — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No